CLINICAL TRIAL: NCT05189795
Title: The Construction and Demonstration of Physical ACtivity Enhancement Scheme (PACES) in Hemodialysis Patients
Brief Title: The Construction of Physical ACtivity Enhancement Scheme (PACES) in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Mei Huang, student, Xi'an Jiaotong University
Other Study IDs: 2021SF-278
Record Dates: First submitted 2021-11-27; First posted 2022-01-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Renal Dialysis; Exercise
Keywords: hemodialysis; physical activity; barriers; benefits
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemodialysis (HD) is the most commonly used renal replacement therapy in patients with end-stage renal disease (ESRD). More than 553,000 ESRD patients in China are currently receiving HD, but the long-term survival rate is low and the mortality rate is as high as 18%, which is significantly associated with low physical activity (PA). Low PA could decrease cardiopulmonary and muscle function, limit the ability to perform activities of daily living, and increase risk of death. The National Kidney Foundation Disease Outcomes Quality Initiative (K/DOQI) recommends PA as cornerstone of ESRD rehabilitation. However, HD patients still live with inactive lifestyle. The investigators' previous study have demonstrated that enhancing PA benefits physical function in HD patients. Therefore, this study intends to establish Physical ACtivity Enhancement Scheme (PACES), that is, to take PACES (measured by pedometers) as the investigation core and motivate patients to PACES.

This study will consists of three distinct parts: 1, 2 and 3. In Part 1, the investigators will conduct research on the PA of HD patients through pedometer and questionnaire, and understand the participants' attitude to PA through a series of questionnaires. In Part 2, the investigators will conduct a semi-structured interview to understand HD patients' attitudes and habits towards PA, as well as recommendations for PACES. In Part 3, the investigators will take the results of Part 1 and 2 as the initial draft of PACES and modify the initial draft through the Delphi method to form the final PACES.

The study aims to develop PACES from the perspective of patients to address the above cognitive factors, making it easier for HD patients to enhance PA.

ELIGIBILITY:
Inclusion Criteria:

* adult (age≥18) with stable ESRD;
* receiving≥3 months HD;
* receiving HD more than 5 times every two weeks;
* volunteer for participating in this investigation.

Exclusion Criteria:

* are unable to do walk on one's own (severe musculoskeletal pain at rest or with minimal activity precluding walking or stationary cycling; unable to sit, stand or walk unassisted, walking devices such as cane or walker allowed);
* have shortness of breath at rest or with activities of daily living (NYHA Class IV);
* have mental disease, disturbance of consciousness and couldn't cooperate with this investigation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This investigation intends to investigate the patients in hemodialysis centers of four hospitals in Xi 'an, and include all patients who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
daily steps (paces) | Within 48 hours of admission to hospital.
  OMRON electronic pedometer (HJ-321) records the participants' daily steps. Participants are instructed to wear the pedometer on their waist for 7 days, and the pedometer is removed only during rest, bathing and swimming.
The Human Activity Profile (HAP) | Within 48 hours of admission to hospital.
  HAP is a questionnaire designed to assess general physical activity. It consists of a list of 94 activities ranked in ascending order of level of energy required to perform each activity. Two scores are available from the HAP: a maximum activity score (MAS), reflective of the most taxing activity a respondent is still perform- ing and an adjusted activity score (AAS), reflective of the respondent's daily activity level. The MAS is the number of the highest ranked activity the respondent is still performing. The AAS is calculated by subtracting from the MAS the number of activities that the respondent has stopped performing that rank below the participants' most metabolically intense activity.
Expectations and challenges of PA enhancement in HD patients | 6 months.
  The outcomes are qualitative information acquired from semi-structured interviews.

SECONDARY OUTCOMES:
Dialysis Patient-perceived Exercise Benefits and Barriers Scale (DPEBBS) | Within 48 hours of admission to hospital.
  The 24-item DPEBBS is used to evaluate participants' perceived benefits and barriers to exercise. The scale consisted of 24 items and 2 open questions, including 12 items of exercise benefits and 12 items of exercise barriers. Total scores ranged from 24 to 96. The higher the score, the more exercise benefits the patients experienced and the fewer factors that prevented them from exercise.
Self-efficacy for exercise scale (SEE) | Within 48 hours of admission to hospital.
  SEE is used to identify the participants' confidence in their ability to exercise, which is a major determinant in the success of changing behavior. The score ranges from 0 to 100, and the higher the score, the higher the level of self-efficacy.
Social support Rating Scale (SSRS) | Within 48 hours of admission to hospital.
  Participants' social support status is measured by the SSRS. The scale has 10 items, including 3 aspects, objective support, subjective support and utilization of social support. The total score is the sum of points for each item. The higher the score is, the higher the degree of social support is. The scale scores range from 12 to 66, with ≤22 being low, 23 to 44 medium, and 45 to 66 high.
Stage of Change Questionnaire | Within 48 hours of admission to hospital.
  The questionnaire identifies the participants' state of readiness to adopt a more active lifestyle according to the Health Action Process Approach.
Kidney Disease Quality of Life (KDQOL-36) | Within 48 hours of admission to hospital.
  KDQOL-36, consisted of the 12-item Short Form Health Survey (SF-12) including the physical component summary (PCS) and the mental component summary (MCS) and 24 disease-specific items which entail 3 subscales: the symptom and problems list, the burden of kidney disease, and the effects of kidney disease, is to evaluate patients' QoL. Scores of each dimension range from 0 to 100 and higher scores represent better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Chunping Ni, doctor, Study Director — Nursing School of the Air Force Medical University
Locations (1):
- Nursing School of the Air Force Medical University, Xi'an, Shaan'xi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang M, Lv A, Yang F, Tang Y, Li Y, Hua Y, Gao J, Ni C. Impacts of cognition of exercise on physical activity participation in hemodialysis patients. Semin Dial. 2023 Sep-Oct;36(5):366-373. doi: 10.1111/sdi.13138. Epub 2023 Jan 3. PMID 36597274

DOCUMENTS (1):
  • Informed Consent Form (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT05189795/ICF_000.pdf